CLINICAL TRIAL: NCT00794417
Title: A Phase 1/2 Study of Aflibercept Administered in Combination With Pemetrexed and Cisplatin in Patients With Advanced Carcinoma
Brief Title: A Study of Aflibercept Administered in Combination With Pemetrexed and Cisplatin in Participants With Advanced Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFT-ST-0708; TCD10767
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Advanced Carcinoma; Non-small Cell Lung Cancer
Keywords: advanced cancer; lung cancer; NSCLC; Non-small Cell Lung Cancer; aflibercept; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — aflibercept; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin (Experimental): Participants received intravenous infusion of aflibercept 6 mg/kg followed by pemetrexed 500 mg/m^2 and then cisplatin 75 mg/m^2 on Day 1 of each 3 week cycle (1 Cycle = 21 Days in this study) until disease progression, unacceptable toxicity, withdrawal of consent or if another study withdrawal criterion has been met.
  Interventions: Drug: Aflibercept; Drug: Pemetrexed; Drug: Cisplatin
- Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin (Experimental): Participants received intravenous infusion of aflibercept 2 milligrams per kilogram (mg/kg) followed by pemetrexed 500 mg/square meter (m^2) and then cisplatin 75 mg/m^2 on Day 1 of each 3 week cycle (1 Cycle = 21 Days in this study) until disease progression, unacceptable toxicity, withdrawal of consent or if another study withdrawal criterion has been met.
  Interventions: Drug: Aflibercept; Drug: Pemetrexed; Drug: Cisplatin
- Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin (Experimental): Participants received intravenous infusion of aflibercept 4 mg/kg followed by pemetrexed 500 mg/m^2 and then cisplatin 75 mg/m^2 on Day 1 of each 3 week cycle (1 Cycle = 21 Days in this study) until disease progression, unacceptable toxicity, withdrawal of consent or if another study withdrawal criterion has been met.
  Interventions: Drug: Aflibercept; Drug: Pemetrexed; Drug: Cisplatin
- Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin (Experimental): Participants received intravenous infusion of aflibercept 6 mg/kg followed by pemetrexed 500 mg/m^2 and then cisplatin 75 mg/m^2 on Day 1 of each 3 week cycle (1 Cycle = 21 Days in this study) for 6 cycles.
  Interventions: Drug: Aflibercept; Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Aflibercept — Administered in combination with the other two interventions via intravenous infusion.
Drug: Pemetrexed — Administered in combination with the other two interventions via intravenous infusion.
  Other Names: Alimta
Drug: Cisplatin — Administered in combination with the other two interventions via intravenous infusion.
  Other Names: Platinol

SUMMARY:
The purpose of the study was to determine whether the combination of aflibercept, pemetrexed and cisplatin is safe and effective in treating non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
The study was conducted in two phases. In phase 1, patients with advanced cancer received different doses of aflibercept in combination with approved doses of pemetrexed and cisplatin. The objective of phase 1 was to determine the safest dose of the combined study medications. This dose was administered to patients with previously untreated NSCLC in phase 2. The phase 2 portion of the study determined if the combination is effective in treating NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of cancer by biopsy (tissue sample)
* Phase 1: patients with advanced or metastatic disease that have failed conventional therapy
* Phase 2: patients with previously untreated NSCLC, excluding squamous cell histology and cavitating lesions
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate renal, liver and bone marrow function.
* Negative pregnancy test (serum or urine) in females of childbearing potential within 7 days of the initial dose of aflibercept
* Ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Institutional Review Board (IRB) approved, signed and dated informed consent form

Exclusion Criteria:

* Prior treatment with study medications
* Untreated, symptomatic, or progressive Central Nervous System cancer and/or spinal cord compression. Patients with treated brain metastases must have been without symptoms for at least 3 months
* Surgery up to 4 weeks prior to the initial administration of aflibercept and/or incomplete wound healing
* Anti-VEGF therapy up to 4 weeks prior to the initial administration of aflibercept (for phase 1 only)
* Chemotherapy up to 4 weeks prior to the initial administration of aflibercept (for phase 1 only)
* Other investigational treatment up to 4 weeks prior to the initial administration of aflibercept
* Any of the following up to 6 months (24 weeks) prior to the initial administration of aflibercept:

  * Severe cardiovascular disease or event
  * Cerebrovascular accident, transient ischemic attack, or moderate to severe peripheral neuropathy
  * Erosive esophagitis or gastritis, infectious or inflammatory bowel disease, and diverticulitis
  * Deep vein thrombosis, pulmonary embolism, or other clotting event
  * Episode(s)of moderate to severe, continuous bleeding
* Breast-feeding or pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-11-30 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2011-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (15):
- United States (14):
  - Arizona Cancer Institute, LLC, Tucson, Arizona
  - University of Arkansas for Medical Science, Little Rock, Arkansas
  - Stanford University Medical Center, Stanford, California
  - Palm Beach Institute of Hematology and Oncology, Boynton Beach, Florida
  - Edward Hines Jr. VA Medical Center, Hines, Illinois
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - UNM Cancer Clinic, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Montefiore Medical Center, The Bronx, New York
  - Presbyterian Hospital Center for Cancer Research, Charlotte, North Carolina
  - Erie Regional Cancer Center, Erie, Pennsylvania
  - Schiffler Cancer Center - Medical Oncology Division, Wheeling, West Virginia
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Diaz-Padilla I, Siu LL, San Pedro-Salcedo M, Razak AR, Colevas AD, Shepherd FA, Leighl NB, Neal JW, Thibault A, Liu L, Lisano J, Gao B, Lawson EB, Wakelee HA. A phase I dose-escalation study of aflibercept administered in combination with pemetrexed and cisplatin in patients with advanced solid tumours. Br J Cancer. 2012 Aug 7;107(4):604-11. doi: 10.1038/bjc.2012.319. Epub 2012 Jul 17. PMID 22805331
- [Result] Chen H, Modiano MR, Neal JW, Brahmer JR, Rigas JR, Jotte RM, Leighl NB, Riess JW, Kuo CJ, Liu L, Gao B, Dicioccio AT, Adjei AA, Wakelee HA. A phase II multicentre study of ziv-aflibercept in combination with cisplatin and pemetrexed in patients with previously untreated advanced/metastatic non-squamous non-small cell lung cancer. Br J Cancer. 2014 Feb 4;110(3):602-8. doi: 10.1038/bjc.2013.735. Epub 2013 Nov 28. PMID 24292447

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of 2 phases: phase 1 and phase 2. A total of 18 participants were enrolled in phase 1 of the study and 42 participants were enrolled in phase 2 of the study. Participants enrolled in phase 1 were not eligible for enrollment in phase 2.
Period: Phase 1: Baseline (Day 1) up to Day 751
Arm/Group | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin
Started | 4 | 7 | 7 | 0
Completed | 1 | 4 | 4 | 0
Not Completed | 3 | 3 | 3 | 0
Not completed — Death | 0 | 0 | 2 | 0
Not completed — Other un-specified | 3 | 3 | 1 | 0
Period: Phase 2: Baseline (Day 421) to Day 972
Arm/Group | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin
Started | 0 (Participants enrolled in phase 1 were not eligible for enrollment in phase 2.) | 0 (Participants enrolled in phase 1 were not eligible for enrollment in phase 2.) | 0 (Participants enrolled in phase 1 were not eligible for enrollment in phase 2.) | 42
Completed | 0 | 0 | 0 | 7
Not Completed | 0 | 0 | 0 | 35
Not completed — Death | 0 | 0 | 0 | 7
Not completed — Physician Decision | 0 | 0 | 0 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4
Not completed — Other unspecified | 0 | 0 | 0 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin | Total
Number analyzed (Participants) | 4 | 7 | 7 | 42 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5 | 23 | 33
  >=65 years | 0 | 6 | 2 | 19 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 19 | 28
  Male | 1 | 3 | 5 | 23 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 2
  White | 3 | 7 | 7 | 36 | 53
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Recommended Dose of Aflibercept for Phase 2
Description: Recommended Dose was defined as the highest combination dose at which fewer than 33 percent (%) of participants experienced dose limiting toxicity during the first cycle of therapy.
Time Frame: Phase 1: Baseline up to 315 Days
Population: Full analysis set (FAS) included all participants who were enrolled and received at least one dose of study drug. Data for this outcome measure has been reported for all participants in single arm.
Measure: Number; unit: mg/kg
Groups:
- Phase 1: All Participants: All participants who received intravenous infusion of aflibercept 2 mg/kg or 4 mg/kg or 6 mg/kg followed by pemetrexed 500 mg/square metere (m^2) and then cisplatin 75 mg/m^2 on Day 1 of each 3 week cycle until disease progression, unacceptable toxicity, withdrawal of consent or if another study withdrawal criterion has been met.
Arm/Group | Phase 1: All Participants
Number analyzed (Participants) | 18
mg/kg | 6

2. Secondary Outcome: Phase 2: Objective Response Rate
Description: Objective response rate was defined as the percentage of participants who achieved complete response (CR) or partial response (PR) as assessed by modified Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking the Baseline sum LD as reference.
Time Frame: Phase 2: Baseline (Day 421) up to end of study (Day 972)
Population: FAS included all participants who were enrolled and received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin
Number analyzed (Participants) | 42
Percentage of Participants | 23.8

3. Secondary Outcome: Phase 2: Progression-free Survival (PFS)
Description: PFS was defined as the time in days from the date of first study drug administration to the date of first documentation of tumor progression or death from any cause, whichever occurs first, as assessed by the modified RECIST. Median time of PFS was estimated using Kaplan-Meier method.
Time Frame: Phase 2: Baseline (Day 421) up to end of study (Day 972)
Population: FAS included all participants who were enrolled and received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin
Number analyzed (Participants) | 42
Days | 149 [130 to 212]

4. Secondary Outcome: Phase 1 and 2: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (for example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) was defined as an adverse event with an onset that occurs after receiving study drug. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: Phase 1: Baseline up to 751 Days; Phase 2: Baseline (Day 421) up to 972 Days
Population: FAS included all participants who were enrolled and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin
Number analyzed (Participants) | 4 | 7 | 7 | 42
Participants | 4 | 7 | 7 | 42

5. Secondary Outcome: Phase 1 and 2: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of Aflibercept
Description: The AUC0-inf was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity.
Time Frame: Phase 1 and 2: Pre-dose up to Day 22 post-dose
Population: FAS included all participants who were enrolled and received at least one dose of study drug. Here "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Day*milligrams per liter (mg/L)
Arm/Group | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin
Number analyzed (Participants) | 4 | 6 | 6 | 7
Day*milligrams per liter (mg/L) | 201 (96.5) | 330 (251) | 442 (152) | 402 (100)

6. Secondary Outcome: Phase 1 and 2: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of Pemetrexed
Description: as for outcome 5
Time Frame: Phase 1 and 2: Pre-dose up to Day 1 post-dose, Day 2 post-dose (only in Phase 1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Hour*milligrams per liter (mg/L)
Arm/Group | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin
Number analyzed (Participants) | 4 | 7 | 7 | 10
Hour*milligrams per liter (mg/L) | 151 (30.0) | 151 (32.5) | 162 (12.6) | 148 (24.3)

7. Secondary Outcome: Phase 1 and 2: Maximum Observed Plasma Concentration (Cmax) of Aflibercept and Pemetrexed
Description: Cmax is the maximum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: Phase 1 and 2: Aflibercept: Pre-dose up to Day 22 post-dose; Pemetrexed: Pre-dose up to Day 1 post-dose, Day 2 post-dose (only in Phase 1)
Population: FAS included all participants who were enrolled and received at least one dose of study drug. Here "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable for specific category.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin
Number analyzed (Participants) | 4 | 7 | 7 | 21
mg/L
  Aflibercept: number analyzed (Participants) | 4 | 6 | 7 | 21
  Aflibercept | 53.6 (7.14) | 68.6 (18.7) | 148 (108) | 104 (26.2)
  Pemetrexed: number analyzed (Participants) | 4 | 7 | 7 | 20
  Pemetrexed | 124 (12.6) | 112 (34.7) | 113 (24.6) | 76.8 (40.5)

8. Secondary Outcome: Phase 1 and 2: Total Body Clearance of Aflibercept
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Phase 1 and 2: Pre-dose up to Day 22 post-dose
Population: FAS included all participants who were enrolled and received at least one dose of study drug. Here "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Liter/Day/kg
Arm/Group | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin
Number analyzed (Participants) | 4 | 6 | 6 | 7
Liter/Day/kg | 0.011 (0.004) | 0.016 (0.007) | 0.016 (0.009) | 0.016 (0.004)

9. Secondary Outcome: Phase 1 and 2: Total Body Clearance of Pemetrexed
Description: as for outcome 8
Time Frame: Phase 1 and 2: Pre-dose up to Day 1 post-dose, Day 2 post-dose (only in Phase 1)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Liter/hour/m^2
Arm/Group | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin
Number analyzed (Participants) | 4 | 7 | 7 | 10
Liter/hour/m^2 | 3.40 (0.59) | 3.47 (0.84) | 3.10 (0.22) | 3.49 (0.76)

10. Secondary Outcome: Phase 1 and 2: Terminal Half-Life (t1/2) of Aflibercept
Description: Terminal half-life was defined as the time required for the plasma concentration of drug to decrease 50 percent in the final stage of its elimination.
Time Frame: Phase 1 and 2: Pre-dose up to Day 22 post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin
Number analyzed (Participants) | 4 | 6 | 6 | 7
Days | 3.16 (0.570) | 5.53 (5.43) | 3.72 (1.04) | 4.62 (1.46)

11. Secondary Outcome: Phase 1 and 2: Terminal Half-Life (t1/2) of Pemetrexed
Description: as for outcome 10
Time Frame: Phase 1 and 2: Pre-dose up to Day 1 post-dose, Day 2 post-dose (only in Phase 1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin
Number analyzed (Participants) | 4 | 7 | 7 | 10
Hours | 1.47 (0.39) | 1.63 (0.22) | 1.73 (0.37) | 1.48 (0.34)

12. Secondary Outcome: Phase 1 and 2: Number of Participants With Positive Anti-drug Antibody (ADA) of Aflibercept
Description: Serum samples were analyzed by a validated electrochemiluminescence immunoassay to detect the presence of ADA.
Time Frame: Phase 1: Baseline up to 315 Days; Phase 2: Baseline (Day 421) up to Day 739
Population: FAS included all participants who were enrolled and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin
Number analyzed (Participants) | 4 | 7 | 7 | 42
Participants | 0 | 0 | 1 | 2

13. Secondary Outcome: Phase 1 and 2: Number of Participants With All Grade Glucose Abnormalities
Time Frame: Phase 1: Baseline up to 751 Days; Phase 2: Baseline (Day 421) up to 972 Days
Population: FAS included all participants who were enrolled and received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin
Number analyzed (Participants) | 4 | 7 | 7 | 42
Participants
  Hyperglycemia (Non-Fasting) | 4 | 6 | 7 | 37
  Hyperglycemia (Fasting) | 1 | 3 | 6 | 6
  Hypoglycemia (Non-Fasting) | 0 | 0 | 0 | 5
  Hypoglycemia (Fasting) | 0 | 0 | 0 | 0

14. Secondary Outcome: Phase 1 and 2: Number of Participants With All Grade Hematology Abnormalities
Time Frame: Phase 1: Baseline up to 751 Days; Phase 2: Baseline (Day 421) up to 972 Days
Population: FAS included all participants who were enrolled and received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin
Number analyzed (Participants) | 4 | 7 | 7 | 42
Participants
  Absolute Neutrophil Count (ANC) | 2 | 4 | 7 | 13
  Hemoglobin | 3 | 7 | 6 | 16
  Platelet Count | 2 | 4 | 2 | 8

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to 751 Days for Phase 1 and 972 Days for Phase 2 regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent adverse events (TEAEs). A TEAE is an AE that either begins on or after study drug administration or is a pre-existing condition that worsens on or after study drug administration.
Arm/Group | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/7 | 1/7 | 5/42
Serious Adverse Events (participants affected / at risk) | 1/4 | 5/7 | 3/7 | 16/42
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7 | 7/7 | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin (N=4) | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin (N=7) | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin (N=7) | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin (N=42)
CHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYDROPNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DISEASE PROGRESSION (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
METASTATIC PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
GINGIVAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
METASTATIC PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
REVERSIBLE POSTERIOR LEUKOENCEPHALOPATHY SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPEECH DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Aflibercept 2 mg/kg and Pemetrexed and Cisplatin (N=4) | Phase 1: Aflibercept 4 mg/kg and Pemetrexed and Cisplatin (N=7) | Phase 1: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin (N=7) | Phase 2: Aflibercept 6 mg/kg and Pemetrexed and Cisplatin (N=42)
NAUSEA (Gastrointestinal disorders) | 4 (6) | 5 (6) | 6 (11) | 28 (42)
VOMITING (Gastrointestinal disorders) | 4 (4) | 4 (4) | 4 (6) | 10 (19)
CONSTIPATION (Gastrointestinal disorders) | 3 (4) | 3 (4) | 6 (10) | 22 (29)
DIARRHOEA (Gastrointestinal disorders) | 2 (3) | 2 (4) | 4 (7) | 16 (27)
STOMATITIS (Gastrointestinal disorders) | 1 (2) | 3 (4) | 1 (6) | 15 (18)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 3 (4) | 1 (1) | 12 (14)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (2) | 2 (2) | 1 (1) | 2 (2)
ODYNOPHAGIA (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASCITES (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
GINGIVAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RETCHING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
OROPHARYNGEAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
FATIGUE (General disorders) | 4 (12) | 6 (12) | 6 (29) | 28 (40)
FEELING ABNORMAL (General disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 2 (3) | 1 (1) | 0 (0) | 3 (3)
OEDEMA PERIPHERAL (General disorders) | 2 (3) | 0 (0) | 1 (1) | 5 (6)
MUCOSAL INFLAMMATION (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
XEROSIS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
INFUSION SITE WARMTH (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOCALISED OEDEMA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TEMPERATURE INTOLERANCE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 3 (5) | 3 (8) | 2 (2)
GAIT DISTURBANCE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
INJECTION SITE REACTION (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHILLS (General disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (11)
PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
CYST (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 4 (4) | 1 (1) | 4 (4) | 15 (16)
HEADACHE (Nervous system disorders) | 3 (4) | 1 (1) | 4 (8) | 13 (18)
DIZZINESS (Nervous system disorders) | 1 (1) | 2 (4) | 4 (4) | 6 (6)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 0 (0) | 2 (4) | 4 (5)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
HYPERSOMNIA (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
SINUS HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CLONUS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
INSOMNIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
ANOREXIA (Metabolism and nutrition disorders) | 3 (3) | 4 (9) | 5 (12) | 13 (14)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 0 (0) | 6 (12)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 12 (19)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 1 (1) | 4 (5)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 7 (8)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (14)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
WEIGHT LOSS POOR (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (15)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (13)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (10)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (9)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 4 (4) | 14 (14)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5) | 3 (3) | 7 (7)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (4) | 2 (2) | 0 (0)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (4) | 1 (1) | 5 (6)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 5 (5) | 11 (12)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 7 (9)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 6 (6)
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
HYPOVENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NASAL ULCER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RHONCHI (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
HYPERTENSION (Vascular disorders) | 2 (6) | 3 (3) | 5 (8) | 22 (34)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (4) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
MUSCLE TWITCHING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (4) | 5 (7)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 2 (2) | 5 (5)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 2 (7) | 5 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (5)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 2 (3)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (7)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 4 (4)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
ORAL HERPES (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HERPES VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN ODOUR ABNORMAL (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SWELLING FACE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 4 (4)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAIR TEXTURE ABNORMAL (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VISION BLURRED (Eye disorders) | 2 (2) | 0 (0) | 2 (3) | 4 (4)
EYE IRRITATION (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
PHOTOPHOBIA (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DRY EYE (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
MYODESOPSIA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 0 (0) | 5 (18)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 7 (11)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 7 (19)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (6)
TINNITUS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (4) | 3 (3)
DEAFNESS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AURICULAR SWELLING (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EAR CANAL STENOSIS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOACUSIS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
HEART RATE DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 2 (5) | 4 (12) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (5) | 2 (3)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (3) | 2 (3)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (6) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 8 (21)
BLADDER DISCOMFORT (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 14 (21)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
AMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (5)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
ABNORMAL DREAMS (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HALLUCINATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOSS OF LIBIDO (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
SCRATCH (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OPEN WOUND (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.